CLINICAL TRIAL: NCT04245020
Title: An Open Label Randomised Control Trial Comparing Three Methods of Outpatient Follow up After Surgical Admission in Connolly Hospital Blanchardstown; Text Message, Phone Call and In-person Appointment
Brief Title: A Study Comparing Three Methods of Outpatient Follow up After Surgical Admission; Text Message, Phone Call and In-person Appointment
Acronym: ISOTOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connolly Hospital Blanchardstown (Other)
Responsible Party: Principal Investigator, Paul Cromwell, General Surgery SpR, Connolly Hospital Blanchardstown
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISOTOPE
Record Dates: First submitted 2019-09-15; First posted 2020-01-28 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Outpatients; Virtual Clinic; Text Messaging; General Surgery
Keywords: Randomised control trial; Virtual clinic; Text messaging; General surgery; Outpatients; Satisfaction; Telemedicine
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Text Message (Active Comparator): Patients will be followed up with a series of text messages at 6-8 weeks
  Interventions: Other: Text message follow up
- Telephone (Active Comparator): Patients will be followed with a telephone conversation at 6-8 weeks
  Interventions: Other: Telephone follow up
- In person (Active Comparator): Patients will be followed in person in the Outpatient department at 6-8 weeks
  Interventions: Other: In person follow up

INTERVENTIONS:
Other: Text message follow up — A text message will be sent to the patient 6-8 weeks following discharge
  Arms: Text Message
Other: Telephone follow up — The patient will be followed up at 6-8 weeks following discharge with a telephone call
  Arms: Telephone
Other: In person follow up — The patient will be followed up at 6-8 weeks following discharge in person in the outpatient department
  Arms: In person

SUMMARY:
This study compares three different methods of outpatient follow up after surgical admission to Connolly Hospital Blanchardstown. The three arms of the study are text message, telephone call or in-person outpatient follow up. Data will be collected to identify complications identified in each arm along with the rate of non-response to the follow up methods and the level of satisfaction with the method. Willingness to use a telemedicine app in the future will also be evaluated through satisfaction survey.

DETAILED DESCRIPTION:
This is a non-blinded, single centre open randomised control trial of the outpatient follow up method following surgical admission to Connolly Hospital Blanchardstown.

All eligible patients will be randomised into three arms, text message, telephone or in-person follow up. The follow up will be carried out at 6-8 weeks following discharge. The rate of complications, the non-response rate and the level of satisfaction will be compared between the three groups.

Willingness to use a telemedicine app in the future in place of an in-person follow up will also be measured by patient satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients admitted either as an emergency or for an elective procedure
* 16 years or older

Exclusion Criteria:

* Did not consent or cannot give consent
* Age less than 16
* No smartphone
* Further follow up required for treatment of further investigation
* Diagnosis or suspected diagnosis of malignancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Complications that require further follow up | 6-8 weeks
  Complications are identified by patient record and follow up method selected

SECONDARY OUTCOMES:
Satisfaction in follow up | 8-10 weeks
  A questionnaire will assess how happy based on a survey patients were with their follow up method. The CSQ 8 score will be used along with a previously published questionnaire from this institiution. In the CSQ-8 questionnaire a higher score indicates more satisfaction.
Willingness to use a virtual clinic app in the future | 8-10 weeks
  A questionnaire will assess patients preference in further follow up, specifically are patients happy to use a telemedicine based app. (answer no definitely not, no not really, yes generally, yes definitely.
Follow up preference | 8-10 weeks
  Preferred follow up method will be identified by above patient questionnaire (text, phone or OPD)
Lost to follow up | 6-8 weeks
  number of patients that are lost to follow up per follow up method
Further procedures arranged | 8-10 weeks
  number of patients who have an additional procedure arranged which will be identified in the medical record

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Cromwell, BM BS BA MRCS, Principal Investigator — Department of Surgery, Connolly Hospital Blanchardstown, Dublin 15; Thomas N Walsh, MD MCh FRCSI, Study Chair — Department of Surgery, Connolly Hospital Blanchardstown, Dublin 15
Locations (1):
- Connolly Hospital Blanchardstown, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided
All data will be shared with other researchers if requested